CLINICAL TRIAL: NCT00216086
Title: A Phase II Trial of Preoperative Capecitabine Plus Irinotecan Followed by Combined Modality Capecitabine and Radiation for Locally Advanced Rectal Cancer: Hoosier Oncology Group GI03-53
Brief Title: Capecitabine + Irinotecan Followed by Combined Modality Capecitabine and Radiation in Locally Advanced Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Gabi Chiorean, MD (Other)
Collaborators: Pfizer (Industry); Roche Pharma AG (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Gabi Chiorean, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GI03-53
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Irinotecan; Neoadjuvant Therapy; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): * Irinotecan 200 mg/m2 IV, day 1
  * Capecitabine 1000* mg/m2 po bid day 1-14; repeat every three weeks for two cycles
    * For calculated creatinine clearance of 30-50 mL/min or patients > 70 years old, capecitabine starting dose is 825 mg/m2 po bid
  * EUS
  * Neoadjuvant Chemotherapy
  * Preoperative Radiation
  * Surgery
  * Adjuvant Chemotherapy (at discretion of treating physician)
  Interventions: Drug: Capecitabine; Drug: Irinotecan; Procedure: EUS; Drug: Neoadjuvant Chemotherapy; Procedure: Preoperative Radiation; Procedure: Surgery; Procedure: Adjuvant Chemotherapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000* mg/m2 po bid day 1-14; repeat every three weeks for two cycles
  *For calculated creatinine clearance of 30-50 mL/min or patients > 70 years old, capecitabine starting dose is 825 mg/m2 po bid
  Other Names: Xeloda
Drug: Irinotecan — Irinotecan 200 mg/m2 IV, day 1
  Other Names: Camptosar
Procedure: EUS — biopsy per EUS
Drug: Neoadjuvant Chemotherapy — * Irinotecan 200 mg/m2 IV, day 1
  * Capecitabine 1000 mg/m2 po bid day 1-14; repeat every three weeks for two cycles
  Other Names: Camptosar; Xeloda
Procedure: Preoperative Radiation — Pelvic XRT 45 Gy/1.8 GY/fx/qd+5/4 Gy/1.8 Gy/fx/qd for T3+9 Gy/1.8/Gy/fx/qd for T4
Procedure: Surgery — Surgery within 8 weeks following chemoradiotherapy
Procedure: Adjuvant Chemotherapy — Adjuvant chemotherapy at investigator's discretion

SUMMARY:
Preoperative induction chemotherapy has been successfully used in a variety of malignancies and provides several advantages over postoperative therapy. Combination of 5-FU/Leucovorin/CPT-11 has demonstrated significantly better response rate than 5-FU/Leucovorin alone. Replacing 5-FU with oral capecitabine in combination with CPT-11 has emerged as a potentially more effective, safe and convenient treatment option for metastatic colorectal cancer. Capecitabine is also well tolerated in concurrent treatment with radiation. Recent data has shown that preoperative radiation appears to be significantly more effective in increasing resectability rates.

This trial will investigate the activity of capecitabine and CPT-11 combination in the preoperative setting followed by chemoradiation with capecitabine in locally advanced rectal cancer to improve response and decrease local recurrence. We will also study whether TS, TP, DPD and carboxyesterase expressions correlate with the objective response rate with this chemotherapy and chemoradiation regimen.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Biopsy per EUS

* Irinotecan 200 mg/m2 IV, day 1
* Capecitabine 1000* mg/m2 PO BID day 1-14 Repeat every three weeks for two cycles* For calculated creatinine clearance of 30-50 mL/min or patients > 70years old, capecitabine starting dose is 825 mg/m2 PO BID

Beginning at week 7 or following recovery from chemotherapy:

* Pelvic XRT 45 Gy/1.8 Gy/fx/qd+5.4 Gy/1.8 Gy/fx/qd for T3+9 Gy/1.8 Gy/fx/qd for T4
* Capecitabine 825* mg/m2 PO BID, 5 days/week, throughout XRT* For calculated creatinine clearance of 30-50 mL/min or patients > 70years old, capecitabine starting dose is 650 mg/m2 PO BID
* Surgery within 8weeks following chemoradiotherapy
* Adjuvant Chemotherapy at investigator's discretion

ECOG performance status 0 or 1

Hematopoietic:·

* ANC count >1,500 mm3·
* Platelets > 100,000/mm3·
* Hemoglobin > 9g/dL
* Prothrombin time (PT)/INR or PTT < 1.25 times upper limit of normal;

Hepatic:·

* Bilirubin <1.5 times upper limit of normal
* Alanine Transaminase (ALT) or Aspartate Transaminase (AST) <2.5 times the upper limit of normal

Renal:·

* Adequate renal function by calculated creatinine clearance > 30 mL/min (by Cockroft and Gault)

Cardiovascular:·

* No congestive heart failure requiring therapy or NYHA class II or greater or active angina or known myocardial infarction within 12 months prior to study

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum < 15 cm from the anal verge without evidence of distant metastasis·
* Measurable disease. ·
* Either mobile cancers (with clinical stage T3 or T4 by endorectal ultrasound) or fixed cancer (defined as clinical T4 for this study) on palpation. ·
* Malignant disease may not extend to the anal canal (across the dentate line)

Exclusion Criteria:

* No prior chemotherapy or radiation therapy to the pelvis.
* Patients with clinical stage T 1-2, N0 rectal cancer who are candidates for primary resection are not eligible·
* No synchronous colonic cancer unless the synchronous tumor is Tis or T1 and has been completely resected·
* Patients must not be taking warfarin·
* No prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-Fluorouracil or known DPD deficiency.·
* No known existing uncontrolled coagulopathy·
* Negative pregnancy test·
* No current breastfeeding·
* No serious concomitant systemic disorders incompatible with the study· No prior malignancies with the exception of curatively treated basal or squamous carcinoma of the skin, carcinoma in-situ of the cervix, or any other cancer for which the patient has been disease-free for < 5 years.·
* Patients must not be treated with any of the following while on protocol therapy or within 28 days prior to beginning protocol therapy: sorivudine, brivudine, cimetidine, allopurinol.
* Patients on dilantin must have regular monitoring of dilantin levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Gabriela Chiorean, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (9):
- United States (9):
  - Elkhart Clinic, Elkhart, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiorean EG, Sanghani S, Schiel MA, Yu M, Burns M, Tong Y, Hinkle DT, Coleman N, Robb B, LeBlanc J, Clark R, Bufill J, Curie C, Loehrer PJ, Cardenes H. Phase II and gene expression analysis trial of neoadjuvant capecitabine plus irinotecan followed by capecitabine-based chemoradiotherapy for locally advanced rectal cancer: Hoosier Oncology Group GI03-53. Cancer Chemother Pharmacol. 2012 Jul;70(1):25-32. doi: 10.1007/s00280-012-1883-1. Epub 2012 May 18. PMID 22610353
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group Assignment: Irinotecan 200 mg/m2 IV, day 1 Capecitabine 1000* mg/m2 po bid day 1-14; repeat every three weeks for two cycles *For calculated creatinine clearance of 30-50 mL/min or patients > 70 years old, capecitabine starting dose is 825 mg/m2 po bid
  Capecitabine: Capecitabine 1000* mg/m2 po bid day 1-14; repeat every three weeks for two cycles
  *For calculated creatinine clearance of 30-50 mL/min or patients > 70 years old, capecitabine starting dose is 825 mg/m2 po bid
  Irinotecan: Irinotecan 200 mg/m2 IV, day 1
  EUS: biopsy per EUS
  Neoadjuvant Chemotherapy: Irinotecan 200 mg/m2 IV, day 1 Capecitabine 1000 mg/m2 po bid day 1-14; repeat every three weeks for two cycles
  Preoperative Radiation: Pelvic XRT 45 Gy/1.8 GY/fx/qd+5/4 Gy/1.8 Gy/fx/qd for T3+9 Gy/1.8/Gy/fx/qd for T4
  Surgery: Surgery within 8 weeks following chemoradiotherapy
  Adjuvant Chemotherapy: Adjuvant chemotherapy at investigator's discretion
Period: Overall Study
Arm/Group | Single Group Assignment
Started | 22
Completed | 18
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Diagnosis of Metastatic Disease | 1
Not completed — Social Reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 54 [36 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    0 | 7
    1 | 15
Tumor Node Metastatis (TNM) Stage [Number; unit: participants] — Tumor Node Metastasis (TNM) Staging. This system classifies tumors by size and extent of the primary tumor (T), involvement of regional lymph nodes (N), and the presence or absence of distant metastases (M) T0=No evidence of primary tumor, Tis=Carcinoma in situ, and T1, T2, T3, T4=Increasing size and/or local extension of the primary tumor, TX=Not assessed N0=No Regional lymph node metastases, N1, N2, N3=Increasing number or extent of regional lymph node involvement, NX=not assessed M0=No distant metastases, M1=Distant metastases present
  participants
    T2 | 1
    T3 | 19
    T4 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: · To determine the pathological response rate of preoperative chemotherapy with capecitabine and irinotecan followed by combined modality chemoradiation with capecitabine in patients with locally advanced rectal cancer.
  Pathological response was defined in the protocol as the proportion of complete (pCR) and non-complete pathological response (pNCR) among all evaluable patients.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 18
percentage of patients
  pCR | 33 [13 to 59]
  pNCR | 56 [31 to 78]

2. Secondary Outcome: Local and Distant Disease Recurrence Rates
Description: To determine the rates of local and distant disease recurrence after treatment.
Time Frame: 36 months
Measure: Number; unit: percentage of particpants
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 18
percentage of particpants
  metastatic disease recurrence | 22
  locally recurrence | 0

3. Secondary Outcome: Rate of Clinical Response
Description: To determine the rate of clinical response following induction chemotherapy with capecitabine and irinotecan, and also the overall clinical response after the completion of chemoradiation with capecitabine.
Time Frame: 36 months
Population: Data for this secondary objective was not captured or analyzed due to the withdrawal of funding and subsequent termination of the study.
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 0

4. Secondary Outcome: Disease-Free Survival
Description: The three year rate of Disease-Free Survival
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 18
percentage | 75.5 [39.7 to 91.8]

ADVERSE EVENTS:
Arm/Group | Single Group Assignment
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group Assignment (N=22)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EDEMA: HEAD AND NECK (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
HYPOTENSION (Cardiac disorders) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group Assignment (N=22)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 9 (13)
APNEA (Psychiatric disorders) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 7 (7)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 18 (32)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 4 (7)
EDEMA: LIMB (Blood and lymphatic system disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 17 (25)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 3 (3)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 3 (4)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 13 (14)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 6 (6)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 4 (4)
HYPOTENSION (Cardiac disorders) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 3 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / PENIS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / VAGINA (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 9 (10)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 4 (4)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 6 (6)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ANUS (Surgical and medical procedures) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 2 (2)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / PHARYNX (General disorders) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / RECTUM (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 16 (22)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 4 (4)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 4 (5)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 4 (4)
PAIN / ANUS (Gastrointestinal disorders) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PAIN / BUTTOCK (General disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / HEAD/HEADACHE (General disorders) | 1 (1)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 7 (8)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1)
PAIN / VAGINA (Reproductive system and breast disorders) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 5 (5)
PLATELETS (Blood and lymphatic system disorders) | 2 (2)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 4 (4)
PROCTITIS (Gastrointestinal disorders) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
PULMONARY HYPERTENSION (Cardiac disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / CHEMORADIATION (Skin and subcutaneous tissue disorders) | 4 (5)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / RADIATION (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 3 (3)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 1 (2)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Psychiatric disorders) | 2 (2)
SWEATING (DIAPHORESIS) (General disorders) | 2 (2)
SYNDROMES - OTHER (SPECIFY, __) (General disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 4 (4)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 7 (9)
WEIGHT LOSS (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No